CLINICAL TRIAL: NCT07098884
Title: Artificial Intelligence for Pathology Diagnosis and Prognosis Prediction of Lung Nodule Using Smartphone Photos
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SPAI
Record Dates: First submitted 2025-07-03; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Artificial Intelligence; Lung Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: AI model — AI model developed by smartphone photos of resected tumor specimens

SUMMARY:
The current study aims to develop and validate a deep learning signature for diagnosing pathology and predicting prognosis of lung nodule using smartphone photos of resected tumor specimens.

ELIGIBILITY:
Inclusion Criteria: (1) Participants scheduled for surgery for radiological finding of pulmonary lesions from the preoperative thin-section CT scans; (2) Age ranging from 20-75 years.

Exclusion Criteria: (1) Participants with incomplete clinical information; (2) Participants who have received anti-tumor therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving surgery for lung nodule
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve | From enrollment to the end of the study, assessed up to 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Individual participant data involve patient privacy and requires strict data protection measures